CLINICAL TRIAL: NCT00743106
Title: The Effect of Fenoldopam on Renal Function in Solitary Partial Nephrectomy Surgery
Brief Title: The Effect of Fenoldopam in Solitary Partial Nephrectomy Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Executive committee determined to close study after interim analysis.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5508
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Partial Nephrectomy
Keywords: nephrectomy; fenoldopam; atrophic minimally functioning kidney
MeSH Terms: interventions — Fenoldopam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Placebo (0.9% Nacl)infusion beginning during surgery and lasting for up to 24 hours
  Interventions: Drug: Placebo
- Fenoldopam Comparator (Active Comparator): Fenoldopam (0.1 ~g/kg/min)infusion will commence after placing the patient in a lateral/flex position during the operation. The infusion will continue for a total of 24 hours.
  Interventions: Drug: Fenoldopam

INTERVENTIONS:
Drug: Fenoldopam — Fenoldopam (0.1 ~g/kg/min)started during surgery and lasting for a total of 24 hours
  Arms: Fenoldopam Comparator
Drug: Placebo — Placebo infusion(0.9% Nacl) beginning during surgery and lasting for up 24 hours post surgery
  Arms: Placebo Comparator

SUMMARY:
This trial will study the effects of fenoldopam on renal function in patients who have a single kidney undergoing surgery to remove part of that kidney secondary to renal cell carcinoma. The investigators will monitor and evaluate throughout the perioperative course the kidney function. Normally kidney function is predicted to show a worsening followed by an improvement after surgery.

The investigators want to specifically identify if the use of fenoldopam lessens the injury to the kidney with this surgery.

DETAILED DESCRIPTION:
Prospective, randomized, blinded study-dividing patients into one of two groups: fenoldopam or placebo. The infusion will commence after placing the patient in a lateral/flex position during the operation. The infusion will continue for a total of 24 hours.Study time period will be approximately six weeks from the date of surgery. Specifically, the following pre- and post operative laboratory results will be recorded if available: . Basic metabolic panel - pre-op, post op days 1, 2, 3, 4, and 6 weeks

* Serum osmolality, urine osmolality, urine sodium - pre-op, post op days 1, 3
* Glomerular filtration rate - pre-op, post op days 1, 3, and 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a solitary kidney and present for a partial nephrectomy
* Patients who have one atrophic minimally functioning kidney and present for partial nephrectomy on the other kidney

Exclusion Criteria:

* History of current renal disease beyond the diagnosis of renal malignancy
* Insulin dependent diabetes mellitus, myocardial infarction without subsequent coronary artery bypass or angioplasty
* History of congestive heart failure, renovascular occlusion greater than 45 minutes or less than 15 minutes, greater than one half of the solitary kidney resected
* A major perioperative complication that would potentially affect postoperative renal function (myocardial infarction, congestive heart failure, pulmonary embolus, massive hemorrhage and hypotension, ureteral obstruction or vascular thrombosis), and evidence of nephrotoxicity due to antibiotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome O'Hara, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — Cleveland Clnic
Locations (1):
- Cleveland Clnic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (0.9% Nacl)infusion beginning during surgery and lasting for up to 24 hours
  Placebo: Placebo infusion(0.9% Nacl) beginning during surgery and lasting for up 24 hours post surgery
- Fenoldopam: Fenoldopam (0.1 ~g/kg/min)infusion will commence after placing the patient in a lateral/flex position during the operation. The infusion will continue for a total of 24 hours.
  Fenoldopam: Fenoldopam (0.1 ~g/kg/min)started during surgery and lasting for a total of 24 hours
Period: Overall Study
Arm/Group | Placebo | Fenoldopam
Started | 42 | 48
Completed | 34 | 43
Not Completed | 8 | 5
Not completed — Met intraoperative exclusion criterion | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fenoldopam | Total
Number analyzed (Participants) | 34 | 43 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9) | 59 (10) | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 29 | 33 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31 | 42 | 73
  Others | 3 | 1 | 4
GFR [Mean (Standard Deviation); unit: mL/min] | 59 (19) | 59 (19) | 59 (19)
creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1.2 [1.0 to 1.4] | 1.2 [1.0 to 1.4] | 1.2 [1.0 to 1.4]

OUTCOME MEASURES:

1. Primary Outcome: Glomerular Filtration Rate (GFR) Percentage of Change From Baseline
Description: Our intended primary analysis was to assess the effect of fenoldopam vs placebo on the GFR at post-operative day (POD) 3 with an analysis of covariance adjusting for the baseline GFR. However, because the intervention-by-baseline GFR interaction using GFR at POD 3 as the outcome was significant (P ¼ .006), the analysis of covariance was not valid. We, therefore, used the GFR percentage of change from baseline to POD 3 as the primary outcome.
Time Frame: percentage of change from baseline to post-operatively day 3
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Fenoldopam
Number analyzed (Participants) | 34 | 43
percentage change | -39 (28) | -28 (38)
Statistical Analysis 1: Comparison: Placebo vs Fenoldopam; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -11, 95% CI 2-sided [-31 to 9] — The mean decrease in GFR was an estimated 11% less for fenoldopam than for placebo (interim-adjusted 95% confidence interval 9% more, 31% less)

2. Secondary Outcome: Postoperative Creatinine (mg/dL)
Description: assessed the effect of fenoldopam on creatinine over time (immediately postoperatively and on postoperative day 1, 2, 3, 4)
Time Frame: "immediately postoperative, postoperative day 1, postoperative day 2, postoperative day 3, postoperative day 4"
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Fenoldopam
Number analyzed (Participants) | 34 | 43
mg/dL
  immediately postoperative | 1.44 (0.07) | 1.37 (0.06)
  postoperative day 1 | 2.14 (0.11) | 2.04 (0.12)
  postoperative day 2 | 2.66 (0.23) | 2.38 (0.19)
  postoperative day 3 | 2.65 (0.25) | 2.46 (0.25)
  postoperative day 4 | 2.76 (0.30) | 2.61 (0.33)
Statistical Analysis 1: Comparison: Placebo vs Fenoldopam; We assessed the effect of fenoldopam on creatinine over time (immediately postoperatively and on PODs 1-4). A linear mixed effects model was used to assess the main effect of fenoldopam on the postoperative log-transformed (base 2) serum creatinine, adjusting for baseline serum creatinine; Test type: Superiority; p = 0.78, Mixed Models Analysis; ratio of geometric mean = 0.98, 95% CI 2-sided [0.79 to 1.19]

ADVERSE EVENTS:
Arm/Group | Placebo | Fenoldopam
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/42
Other Adverse Events (participants affected / at risk) | 0/34 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No